CLINICAL TRIAL: NCT02333149
Title: Melatonin in Youth: N-of-1 Trials in a Stimulant-treated Attention Deficit Hyperactivity Disorder (ADHD) Population
Acronym: MYNAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Issues surrounding the current COVID-19 pandemic.
Sponsor: University of Alberta (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00022025
Record Dates: First submitted 2014-12-16; First posted 2015-01-07 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Initial Insomnia
Keywords: Melatonin
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Dietary supplement: Melatonin 3 mg or 6 mg
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Drug: Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Children <40 kg will take one tablet, melatonin 3 mg, oral, 30 - 60 minutes prior to bedtime.
  Children ≥40 kg will take two tablets, melatonin 3 mg, oral, 30-60 minutes prior to bedtime.
  Arms: Melatonin
Drug: Placebo — Placebo frequency and volume are identical to the experimental arm
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, triple-blind, placebo-controlled parallel-group trial, in which each participant is offered an N-of-1 trial. The purpose of this study is to assess the efficacy and safety of melatonin (3 mg or 6 mg) compared with placebo for initial insomnia in children with attention-deficit disorder.

ELIGIBILITY:
Inclusion Criteria:

* School-aged children and adolescents between the ages of 6 to 17 years
* Confirmed diagnosis of ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)

Exclusion Criteria:

* Co-morbid psychiatric/neurological diagnoses that may affect sleep
* Co-morbid seizure disorder
* Co-morbid sleep disorder
* Concurrent use of immunosuppressive drugs, blood pressure drugs, selective serotonin re-uptake inhibitors or anticoagulant drugs;
* Pregnancy or breastfeeding

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Mean change in sleep onset latency (minutes) | Daily, up to 6 weeks
  The mean change in sleep onset latency will be measured using sleep diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Sunita Vohra, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Punja S, Nikles CJ, Senior H, Mitchell G, Schmid CH, Heussler H, Witmans M, Vohra S. Melatonin in Youth: N-of-1 trials in a stimulant-treated ADHD Population (MYNAP): study protocol for a randomized controlled trial. Trials. 2016 Jul 29;17:375. doi: 10.1186/s13063-016-1499-6. PMID 27473269